CLINICAL TRIAL: NCT01336322
Title: Effects of Treatment With Metformin and/or Sitagliptin on Beta-cell Function and Insulin Resistance in Women With Previous Gestational Diabetes
Brief Title: Metformin and Sitagliptin in Women With Previous Gestational Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pisa (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Prof. Stefano Del Prato, Clinical Resercher, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SITA-previousGDM
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Pre-diabetes
Keywords: beta-cell function; insulin resistance
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Metformin; Sitagliptin Phosphate; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metformin (Active Comparator): Metformin 850 mg bid
  Interventions: Drug: Metformin
- Sitagliptin (Active Comparator): Sitagliptin 100 mg qd
  Interventions: Drug: Sitagliptin
- Sitagliptin+Metformin (Active Comparator): Sitagliptin 100 mg qd plus Metformin 850 mg bid
  Interventions: Drug: Sitagliptin + Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg bid
  Other Names: Glucophage
  Arms: Metformin
Drug: Sitagliptin — Sitagliptin 100 mg qd
  Other Names: januvia
  Arms: Sitagliptin
Drug: Sitagliptin + Metformin — sitagliptin 100mg + metformin 850mg
  Other Names: janumet
  Arms: Sitagliptin+Metformin

SUMMARY:
The goal of the present research is to compare the effects of treatment with metformin and sitagliptin, alone or in association, in women with previous gestational diabetes to evaluate the impact of the two drugs on beta-cell function. The study results may contribute to give a rational approach for future investigations.

DETAILED DESCRIPTION:
A randomized, double blinded study, on 45 women with previous gestational diabetes and impaired glucose tolerance (IGT) or impaired fasting glucose (IFG) to assess the effects of a 4-month treatment with metformin and/or a dipeptidyl peptidase-4 inhibitor (sitagliptin) on beta-cell function and insulin resistance.

At baseline, all women will have a standardized medical history, physical, and laboratory examination. Plasma glucose, insulin, pro-insulin, C-peptide, glucagon, adipokines, pro-inflammatory molecules, and lipid profile will be determined in fasting condition. A 75g OGTT will be performed after an overnight fasting and sample will be drawn at 15, 30, 60, 90 and 120 minutes for plasma glucose, C-peptide, glucagon and GLP-1 determinations. Women with IFG or IGT will be recruited and undergo to a hyperglycemic clamp with arginin bolus at the end of the test. Then the women will be randomized in 3 treatment groups: metformin (850 mg bid), sitagliptin (100 mg qd)or metformin (850 mg bid) + sitagliptin (100 mg qd). After 4-month treatment, the baseline evaluation will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged ≥18 and ≤45 years
* Caucasian race
* History of previous gestational diabetes (in the screening) during pregnancy.
* Female of childbearing potential must use effective contraceptive measures for at last 1 month prior to entry into the study and should continue to use the some contraceptive method during the overall study period
* Written informed consent obtained

Exclusion Criteria:

* Patients diagnosed with type 1 insulin dependent diabetes
* Diagnosis of diabetes in the 75g OGTT performed at entry
* BMI ≤18 or ≥50 Kg/m2
* Chronic impaired renal function
* Impaired liver function as shown by transaminase levels ≥ twice above the upper normal range
* History of hypersensitivity to metformin
* Pregnant or breast-feeding women, or women planning to become pregnant during the study
* Failure to use adequate contraception (Women of current reproductive only)
* Mental condition rending the subject unable to understand the nature, scope and possible consequences of the study
* Any clinically significant major organ system disease
* Patients with underlying concomitant medication requiring a long-term use of drugs potentially acting on glucose metabolism (e.g. corticosteroids, diuretics, beta-adrenergic drugs or others)
* Treatment or likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* History of drug or alcohol abuse within the last 2 years or current addiction to substances of abuse
* Any disease or condition that in the opinion of the investigator may interfere with the completion of the study
* Subjects unlikely to comply with the protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Beta-cell function | 4 months
  Sitagliptin and/or metformin effects on beta-cell function (ISR = Insulin Secretion Rate) evaluated by mathematical model by Mari A. (Am J Physiology 2002)

SECONDARY OUTCOMES:
Insulin resistance | 4 months
  Sitagliptin and/or metformin effects on insulin resistance, evaluated by clamp, HOMA-index and ISI-Method..
Glucose control | 4 months
  Sitagliptin and/or metformin effects on glucose control evaluated by OGTT and HbA1c levels.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Del Prato, MD, Principal Investigator — University of Pisa
Locations (1):
- Department of Endocrinology and Metabolism, University of Pisa, Pisa, Italy